CLINICAL TRIAL: NCT05873660
Title: Multi-centre Cross-sectional Observational Study to Characterize the Prevalence of Overweight and Obesity Among Patients With Established Cardiovascular Disease
Brief Title: A Study to Characterize the Prevalence of Overweight and Obesity Among Patients With Established Cardiovascular Disease
Acronym: POETIC
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: DAS-7537; U1111-1283-8551 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People with established CVD: Adults diagnosed with established CVD, attending routine medical care or follow-up in a cardiology clinic.
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment given

SUMMARY:
The purpose of this observational study is to measure how many people are overweight or obese amongst patients with a diagnosed cardiovascular disease (CVD). The study also aims to characterise the population including the presence of cardiovascular (CV) risk factors in a number of countries across the globe representing different geographies, ethnicities, as well as different healthcare systems.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
2. Adults, age above or equal to 18 years at the time of signing informed consent.
3. Have established CVD and equal to or greater than 1 follow up appointment following an acute event from at least one of the following:

   * Prior myocardial infarction
   * Prior stroke (ischemic or haemorrhagic stroke)
   * Symptomatic peripheral arterial disease (PAD), as evidenced by intermittent claudication with ankle-brachial index (ABI) below 85 (at rest), or peripheral arterial revascularization procedure, or amputation due to atherosclerotic disease

Exclusion Criteria:

1. Previous participation in this study. Participation is defined as having given informed consent in this study
2. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
3. Patients with known congenital heart disease/malformation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adults aged 18 years or older diagnosed with established cardiovascular disease (CVD) and are attending routine medical care or follow-up in a cardiology clinic.
Sampling Method: Non-Probability Sample
Enrollment: 5360 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Overweight and obesity among patients with established CVD pooled across all countries | At the time of patient enrolment (Day 1/Visit 1)
  % of patients

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (5):
- Novo Nordisk Investigational Site, Plainsboro, New Jersey, United States
- Novo Nordisk Investigational Site, São Paulo, Brazil
- Novo Nordisk Investigational Site, Ontario, Canada
- Novo Nordisk Investigational Site, Riyadh, Saudi Arabia
- Novo Nordisk Investigational Site, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
"According to the Novo Nordisk disclosure commitment on novonordisk-trials.com"
URL: http://novonordisk-trials.com